CLINICAL TRIAL: NCT05647252
Title: General Skin and Nasal Decolonization With Octenisan® Set Be-fore and After Elective Orthopedic Surgery in Selected Patients at Elevated Risk for Revision Surgery and Surgical Site Infections
Brief Title: General Decolonization With Octenisan® Set Before Elective Orthopedic Surgery
Acronym: BALGDEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: Industry (Schülke & Mayr AG, Switzerland and Germany) (Unknown)
Responsible Party: Principal Investigator, Ilker Uckay, Prof Dr. med. Ilker Uçkay, Balgrist University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Prov. Wissenschaftsantrag 980
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Elective Surgery; High Risk; Prevention of Surgical Site Infections; Randomized-controlled Trial
Keywords: Body and nasal decolonization; Adult orthopedic surgery; Prevention of Surgical Site Infections; Randomized-controlled trial
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Single-Center, Unblinded, Superiority, Randomized-Controlled Trial (Randomization 1:1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decolonization (Experimental): This study will be performed with an existing "set" manufactured by Schülke & Mayr GmbH. The distribution of octenisan® wash lotion and octenisan® nasal gel in the form of a set (octenisan® set) largely streamlines and facilitates the application and compliance.
  The duration of pre-surgical decolonization is planned to be five days. However, when this pre-surgical time period is too short, the decolonization may also start at least 3 days before surgery and be contin-ued up to 2 days post-surgery.
  During the post-surgery application, the patient will be washed with water and Octenisan® set by their treating nurses. The patient will also return the empty/used set and answer to a short questionnaire during their hospital stay. The study team will recuperate the questionnaire during hospitalization.
  Interventions: Drug: Whole Body and nasal decolonization with octenidin (Octenisan Set); Behavioral: Questionnaire for study participants immediately after the decolonization
- Non-Decolonization (No Intervention): No Decolonization preoperatively

INTERVENTIONS:
Drug: Whole Body and nasal decolonization with octenidin (Octenisan Set) — Octenidin body lotion once a day during the five consecutive days preceding the elective orthopedic surgery, including for the hair.
  Octenidin nasal creme 2-3 times a day in both nasal orifices during the same period
  Arms: Decolonization
Behavioral: Questionnaire for study participants immediately after the decolonization — A questionnaire in GErman language will be handed out to decolonized patients with five questions: Practical difficulties of decolonization, the completeness of scheduled decolonization actions, all adverse events during decolonization and surgery, and two questions regarding the comprehension of the science (indication for decolonization, potential benefit expected in the individual case).
  The questionnaire is handmade and validated by the Investigators.
  Arms: Decolonization

SUMMARY:
The general decolonization of the human body surface by industrial antiseptic agents, before elective surgery is recommended by the World Health Organization (WHO).

A specific randomized-controlled trial specifically among high-risk adult orthopedic patients for infection has not been performed.

In this single-center, prospective, randomized, and controlled superiority trial, which is planned over a period of two years, we target on an orthopedic patient population with an elevated risk for revision surgery and surgical site infections

DETAILED DESCRIPTION:
The general decolonization of the human body surface and, of adjacent pathogen reservoirs such as the nose, by industrial antiseptic agents by the World Health Organization (WHO) for the risk reduction of superficial and deep surgical site infection (SSI). Such a decolonization is regarded as evidence-based in the majority of randomized, and before-after trials, since two decades, although negative studies also exist.

In the orthopedic field, this decolonization is likely to be more effective in elective patients with a proven body colonization of Staphylococcus aureus. The decolonization might be equally efeective in orthopedic patients with an inherent high risk for SSI, for which the majority of future SSI pathogens are skin commensals and S. aureus. These (eventual and future) pathogens of SSI are accessible to the topical agents during the index surgery, if the patients are well instructed and know how to decolonize themselves.

In contrast, this pre-surgical decolonization is only a supplementary measure in the bundle of all combined efforts to prevent revision surgery for infection. Its individual power is limited for young, healthy individuals, for SSIs caused by pathogens from the internal body sites (intestinal, urinary, gynecologic regions), infections acquired on the surgical ward, and in settings with less specialized surgeries and a low volume of surgical experience. Hence, in trials including all patients (or only those carrying S. aureus), the beneficial effect of decolonization can be diluted and provoke an additional costly and cumber-some organizational procedure for the majority of patients with low to moderate SSI risks.

Moreover, many surgical site infections in orthopedic surgery, especially in implant-related surgery, are more due to coagulase-negative staphylococci (CoNS) than for S. aureus.

The hallmark of the CoNS group is S. epidermidis with approximatively 70% resistance (in Switzerland) to standard prophylactic antibiotic agents9, As S. epidermidis is part of the normal human flora, typically the skin flora, and, only becomes pathogenic under certain conditions, a screening for this microorganism is not feasible in common practice,. while the prophylaxis-resistant part of all orthopedic SSI pathogens is at 30-50%.

In this single-center, prospective, randomized, and controlled superiority trial, which is planned over a period of two years, we target on an orthopedic patient population with an elevated risk for revision sur-gery and SSI; inde-pendently of a known body carriage for S. aureus.

This study will be performed with an existing "set" manufactured by Schülke & Mayr GmbH. The "Set" was placed on the market in 2016. The distribution of Octenisan® wash lotion and Octenisan® nasal gel in the form of a set (Octenisan® Set) largely streamlines and facilitates the organizational application and compliance efforts of the study.

Academically and clinically, we will gain insight in the performance of decolonization for a patient population at particular risk of postoperative complications, where every effort to prevent infection is of importance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with an age ≥ 80 years (as considered particularly at risk for SSI)
* Elective orthopedic surgery at the Balgrist
* Chronic immune-suppression (diabetes mellitus, active cancer, cirrhosis CHILD C, renal dialysis, untreated HIV disease, medicamentous immune-suppression equivalent to prednisone ≥ 10 mg/day)
* Elective surgery in ischemic skin (e.g. major amputations)
* Elective surgery on non-diabetic and non-infected ulcerated skin
* Tumor (oncologic) orthopedic surgery
* ASA-Scores 3-4 points

Exclusion Criteria:

* Elective revision orthopedic surgery due to orthopedic infection within the last 12 months in the same area of surgery
* Emergency surgery (defined as planned surgery within the next 48 hours)
* Surgery on infected skin; or surgery under antibiotic treatment for any reason
* "Diabetic foot surgery" (distinct clinical entity; defined as below the ankle)
* Body mass index ≥ 35 kg/m2 (anticipated difficulty of effective decolonization)
* Pregnancy (formality reasons)
* Intolerance or allergy to octenidin and/or ingredients in the Octenisan® set
* Use of any other topical antiseptic agents other than Octenisan® set (except for the duration of one day)
* Patient unable to understand; or under legal guardian for medical decisions
* Anticipated clinical follow-up of less than 6 weeks after surgery.
* ASA-Scores 1-2, and ASA-Score 5 (high risk of postoperative complications)
* Known skin colonization with antibiotic-multiresistant Gram-negative organisms defined by infection control protocols of Switzerland1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1086 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Remission (and inversely surgical site infection) | At 6 weeks after elective orthopedic surgery; or at 1 year for surgeries with orthopedic implants
  Remission is defined as the absence of clinical, anamnestic, radiologic or laboratory signs of infection.
Wound problems after elective surgery | Until week 6 after surgery
  Wound problems (dehiscence, seroma, hematoma, necrosis) occurring after surgery

SECONDARY OUTCOMES:
Unplanned revision surgery for non-infection problems in same time period | At 6 weeks after elective orthopedic surgery; or at 1 year for surgeries with orthopedic implants
  Any revision in the operating theatre due to non-infectious pathologies
Adverse events | At 6 weeks after elective orthopedic surgery; or at 1 year for surgeries with orthopedic implants
  All adverse events during the decolonization and hospitalization periods
Subjective opinion and information on the decolonization | A day within one week after surgery (during the hospitalization)
  Questionnaire with 5 questions only for patients being decolonized

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uçkay, Prof., Principal Investigator — Balgrist University Hospital, Zürich, Switzerland
Locations (2):
- Switzerland (2):
  - Balgrist University Hospital, Zurich, Canton of Zurich
  - Balgrist University Hospital, Zurich

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol will be published separately The results of the study will be a publication
Supporting Information: Study Protocol, CSR
Time Frame: Before and after the study (February 2023 and May 2025)
Access Criteria: Will be published in PubMed

REFERENCES:
- [Result] Uckay I, Hoffmeyer P, Lew D, Pittet D. Prevention of surgical site infections in orthopaedic surgery and bone trauma: state-of-the-art update. J Hosp Infect. 2013 May;84(1):5-12. doi: 10.1016/j.jhin.2012.12.014. Epub 2013 Feb 14. PMID 23414705
- [Result] Tsang STJ, McHugh MP, Guerendiain D, Gwynne P, Boyd J, Laurenson IF, Templeton KE, Lewis S, Simpson AHRW, Walsh TS. Evaluation of Staphylococcus aureus eradication therapy in orthopaedic surgery. J Med Microbiol. 2018 Jun;67(6):893-901. doi: 10.1099/jmm.0.000731. Epub 2018 Apr 19. PMID 29671723
- [Result] Dancer SJ, Christison F, Eslami A, Gregori A, Miller R, Perisamy K, Robertson C, Graves N. Is it worth screening elective orthopaedic patients for carriage of Staphylococcus aureus? A part-retrospective case-control study in a Scottish hospital. BMJ Open. 2016 Sep 6;6(9):e011642. doi: 10.1136/bmjopen-2016-011642. PMID 27601492
- [Result] Prentice HA, Chan PH, Champsi JH, Clutter DS, Maletis GB, Mohan V, Namba RS, Reddy NC, Hinman AD, Fang AS, Yian E, Navarro RA, Norheim EP, Paxton EW. Temporal Trends in Deep Surgical Site Infections After Six Orthopaedic Procedures Over a 12-year Period Within a US-based Healthcare System. J Am Acad Orthop Surg. 2022 Nov 1;30(21):e1391-e1401. doi: 10.5435/JAAOS-D-22-00280. Epub 2022 Sep 7. PMID 36084332
- [Result] Rohrer F, Notzli H, Risch L, Bodmer T, Cottagnoud P, Hermann T, Limacher A, Fankhauser N, Wagner K, Brugger J. Does Preoperative Decolonization Reduce Surgical Site Infections in Elective Orthopaedic Surgery? A Prospective Randomized Controlled Trial. Clin Orthop Relat Res. 2020 Aug;478(8):1790-1800. doi: 10.1097/CORR.0000000000001152. PMID 32058435
- [Derived] Unterfrauner I, Bragatto-Hess N, Studhalter T, Farshad M, Uckay I. General skin and nasal decolonization with octenisan(R) set before and after elective orthopedic surgery in selected patients at elevated risk for revision surgery and surgical site infections-a single-center, unblinded, superiority, randomized controlled trial (BALGDEC trial). Trials. 2024 Jul 8;25(1):461. doi: 10.1186/s13063-024-08173-y. PMID 38978089
- See also: Octenidin Set (Manufacturer's information) — https://www.schuelke.com/wMedia/docs/folder-broschueren/infektionspraevention/schuelke_Praevention-schlaegt-Infektion_Folder-2021.pdf